CLINICAL TRIAL: NCT05744141
Title: The Effect Of Relaxation Exercises Before Cataract Surgery On The Anxiety Level Of Elderly İndividuals
Brief Title: The Effect Of Relaxation Exercises Before Cataract Surgery on Elderly İndividuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Mehmet Ata Demir, principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-48670771-514.99
Record Dates: First submitted 2023-01-10; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Anxiety Level
Keywords: Nursing; Anxiety; Cataract; Relaxation Exercises
MeSH Terms: conditions — Anxiety Disorders; Cataract

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Elderly individuals undergoing relaxation exercises before cataract surgery
  Interventions: Procedure: Relaxation Exercises
- Control Group (No Intervention): Standard care

INTERVENTIONS:
Procedure: Relaxation Exercises — Relaxation exercises consist of voluntary, rhythmic and regular stretching and relaxation of large and small muscle groups until the whole body relaxes. For this exercise application, the "Relaxation Exercises CD" prepared by the Turkish Psychological Association will be used. The CD consists of 30 minutes and relaxation exercises are explained with the sound of a stream accompanied by verbal instructions. This exercise includes rhythmic breathing, muscle relaxation exercises and music (stream sound).
  Arms: Intervention Group

SUMMARY:
The aim of this study was to determine the effect of relaxation exercises applied before cataract surgery on the anxiety level of elderly individuals.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study to determine the effect of relaxation exercises applied before cataract surgery on the anxiety level of elderly individuals. In this context, as a result of the study, it will be concluded about the effect of relaxation exercises applied before cataract surgery on the anxiety level of elderly individuals. It is also aimed to evaluate the effect of relaxation exercises on the preoperative and intraoperative vital signs of elderly individuals and their satisfaction level with the intervention.

Patients who meet the inclusion criteria will be informed about the purpose, content and method of the study during patient admission in the preoperative period, and the sample group (experimental and control) will be formed by obtaining written permission from those who voluntarily agree to participate in the study. The determination of the experimental and control groups will be provided by the random numbers generated by the https://www.randomizer.org/ website. In the sample group (experimental, control), a pilot study will be conducted to evaluate the applicability of the study plan before the implementation (10 experimental, 10 control). In addition, the researcher will explain the application of relaxation exercises within the scope of the research to the patients in the experimental group by accepting the intervention application in the preoperative period.

Formation of the Experimental Group and Interventions:

* First, patients who meet the sample selection criteria will be identified.
* Standardized Mini Mental Test will be administered to patients who are eligible for the study. Patients with a score of 25 and above will be informed about the purpose, content and method of the study by reading the voluntary information form, and those who voluntarily agree to participate in the study and accept the intervention will be included in the study by obtaining verbal and written consent. According to the order of inclusion in the study, the experimental group will be formed from the numbers generated by the https://www.randomizer.org/ website.
* Cataract surgery (phacoemulsification) is usually performed on a daily basis. In this period, firstly, the Information Form will be applied to the patients. Then, preoperative State-Trait Anxiety Inventory and Visual Comparison Scale will be used to determine anxiety levels and vital signs will be evaluated.
* The non-pharmacologic relaxation exercise method will be explained to the patient by the researcher.
* In order to ensure that the 30-minute relaxation exercises can be performed in a comfortable environment, the patient can relax sufficiently, and the patients can make independent decisions in anxiety assessments; care will be taken to ensure that the patient's relatives are not present in the room, the curtain / screen on the patient's bed is closed, there is no urgency for urinary and bowel evacuation, the CD volume is adjusted according to the patient's preference, and the room is quiet and calm. An eye patch will be used during this period to minimize environmental factors.
* Immediately after the intervention, the State Anxiety Inventory and Visual Comparison Scale will be used to measure the individual's anxiety, satisfaction level with the intervention and vital signs will be evaluated.
* When the individual arrives at the operating room, his/her anxiety level and vital signs will be assessed in the waiting room using the State Anxiety Inventory and Visual Comparison Scale. During the operation, vital signs will be monitored on the monitor at 5 minute intervals. The interpretation of vital signs during the operation will be based on the average value of the measurements.

Relaxation Exercises Practice:

* Relaxation exercises consist of voluntary, rhythmic and regular stretching and relaxation of large and small muscle groups until the whole body relaxes. For this exercise application; "Relaxation Exercises CD" prepared by the Turkish Psychologists Association will be used.
* The CD consists of 3 parts. In the first part, the definition and purpose of 10 minutes of deep relaxation and the practices to be considered during the exercise are explained. The second part consists of 30 minutes and explains relaxation exercises with the sound of a stream accompanied by verbal instructions. The 3rd part consists of 30 minutes and includes only relaxation music without instructions.
* In this study, only the second part of the "Relaxation Exercises CD" will be used and it will be applied in the patient's room/bed by the researcher by using a portable VCD/DVD player, adjusting the volume according to the patient's preference, with the help of headphones, taking into account the institutional policy in the preoperative period.

The elderly individuals in the control group will be measured in the same time period as the experimental group without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older,
* At least be able to read and write,
* No problems in terms of hearing, communication (verbal / non-verbal),
* Can communicate in Turkish,
* Mini Mental State Examination Test score of 25 points and above,
* First time cataract surgery under planned topical/local anesthesia.

Exclusion Criteria:

* Lacking cognitive competence,
* Additional eye problems other than cataracts,
* According to the STAI, with additional anxiety problems other than surgery,
* Known psychiatric problems,
* Developing complications during surgery,
* Elderly individuals who have to undergo different anesthesia will not be included in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in STAI-S's Inventory | before and immediately after the relaxation exercise and before surgery (in the operating room waiting room)
  State anxiety (STAI-S) refers to a temporary emotional state related to a specific situation. The STAI -S consists of 20 items. The total score obtained from the scale is between 20-80 and an increase in the score indicates an increase in the level of anxiety. The validity and reliability of the Turkish versions of these instruments have been validated.
STAI-T's Inventory | before the relaxation exercise
  Trait anxiety (STAI-T) represents anxiety as a stable personality character. The STAI -T consists of 20 items. The total score obtained from the scale is between 20-80 and an increase in the score indicates an increase in the level of anxiety. The validity and reliability of the Turkish versions of these instruments have been validated.
Change in Anxiety as Measured by Visual Analog Scale (VAS-A) | before and immediately after the relaxation exercise, in the operating room waiting room and immediately before surgery.
  Measured using the Visual Analogue Scale for Anxiety (VAS-A), on a scale of 0 to 10, in which a higher score means an increased level of anxiety
Change in Blood Pressure | before and immediately after the relaxation exercise, in the operating room waiting room, immediately before surgery and during surgery
  A calibrated digital sphygmomanometer will be used to measure blood pressure. Results will be reported in mmHg.
Change in Pulse Rate | before and immediately after the relaxation exercise, in the operating room waiting room, immediately before surgery and during surgery
  Calibrated digital finger type pulse oximeter will be used for pulse measurement. The results presented as beat per minute.
Change in Respiratory Rate | before and immediately after the relaxation exercise, in the operating room waiting room, immediately before surgery and during surgery
  Respiratory rate per minute. Higher scores mean a worse result.
Change in Peripheral Oxygen Saturation (SpO2) | before and immediately after the relaxation exercise, in the operating room waiting room, immediately before surgery and during surgery
  Calibrated digital finger type pulse oximeter will be used for Peripheral Oxygen Saturation (SpO2). Approaching 100% is considered positive. Higher scores mean a better result.
Change in Body Temperature | before and immediately after the relaxation exercise, in the operating room waiting room (before surgery )
  A calibrated non-contact infrared thermometer will be used to measure body temperature. Results will be reported in Celcius.

SECONDARY OUTCOMES:
Change in Satisfaction as Measured by Visual Analog Scale | before and immediately after the relaxation exercise
  Measured using the Visual Analogue Scale for Satisfaction, on a scale of 0 to 10, in which a higher score means an increased level of satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Beyoğlu Eye Training and Research Hospital, Istanbul, Beyoğlu, Turkey (Türkiye)

REFERENCES:
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Background] Akoğlu, C., & Çelik, G. K. (2020). Katarakt ameliyatı esnasında ağrı ve anksiyete: birinci göz ve ikinci göz cerrahisi arasında karşılaştırma. http://79.123.186.155/handle/20.500.11787/826
- [Background] Aydemir, Ö. ve Köroğlu, E. (2000). Psikiyatri'de Kullanılan Ölçekler. Ankara: Hekimler Yayın Birliği; 153-163.
- [Background] Babacan Yıldız, G., Ur Özçeli k, E., Kolukısa, M., Işık, A.T., Gürsoy, E., Kocaman, G. ve ark. (2015). Eğitimsizler için modifiye edilen Mini Mental Testin (MMSE-E) Türk toplumunda Alzheimer Hastalığı tanısında geçerlik ve güvenilirlilik çalışması. Türk Psikiyatri Dergisi, 26, 1-8.
- [Background] Beaver, H. A. (2019). Cataracts and cataract surgery. Geriatric Ophthalmology: A Competency-Based Approach: Second Edition, 16-26. https://doi.org/10.1007/978-3-030-04019-2_3
- [Background] Chen M, Hill GM, Patrianakos TD, Ku ES, Chen ML. Oral diazepam versus intravenous midazolam for conscious sedation during cataract surgery performed using topical anesthesia. J Cataract Refract Surg. 2015 Feb;41(2):415-21. doi: 10.1016/j.jcrs.2014.06.027. PMID 25661136
- [Background] Choi S, Park SG, Bellan L, Lee HH, Chung SK. Crossover clinical trial of pain relief in cataract surgery. Int Ophthalmol. 2018 Jun;38(3):1027-1033. doi: 10.1007/s10792-017-0554-y. Epub 2017 Jun 20. PMID 28639089
- [Background] Cline ME, Herman J, Shaw ER, Morton RD. Standardization of the visual analogue scale. Nurs Res. 1992 Nov-Dec;41(6):378-80. No abstract available. PMID 1437591
- [Background] Cavdar AU, Yilmaz E, Baydur H. The Effect of Hand Massage Before Cataract Surgery on Patient Anxiety and Comfort: A Randomized Controlled Study. J Perianesth Nurs. 2020 Feb;35(1):54-59. doi: 10.1016/j.jopan.2019.06.012. Epub 2019 Sep 21. PMID 31551136
- [Background] Dahshan D, Kuzbel J, Verma V. A role for music in cataract surgery: a systematic review. Int Ophthalmol. 2021 Dec;41(12):4209-4215. doi: 10.1007/s10792-021-01986-9. Epub 2021 Jul 26. PMID 34312781
- [Background] Facco E, Stellini E, Bacci C, Manani G, Pavan C, Cavallin F, Zanette G. Validation of visual analogue scale for anxiety (VAS-A) in preanesthesia evaluation. Minerva Anestesiol. 2013 Dec;79(12):1389-95. Epub 2013 Jul 9. PMID 23860442
- [Background] Farmahini Farahani M, Noruzi Zamenjani M, Nasiri M, Shamsikhani S, Purfarzad Z, Harorani M. Effects of Extremity Massage on Preoperative Anxiety: A Three-Arm Randomized Controlled Clinical Trial on Phacoemulsification Candidates. J Perianesth Nurs. 2020 Jun;35(3):277-282. doi: 10.1016/j.jopan.2019.10.010. Epub 2020 Feb 10. PMID 32057627
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gadegone, A., Daigavane, S., & Walavalkar, R. (2021). Effect of Music on Blood Pressure and Heart Rate in Patients Undergoing Cataract Extraction Surgery. Original Research Article J Evolution Med Dent Sci, 10. https://doi.org/10.14260/jemds/2021/309
- [Background] Giannaccare G, Bernabei F, Pellegrini M, Guaraldi F, Turchi F, Torrazza C, Senni C, Scotto R, Sindaco D, Di Cello L, Versura P, Scorcia V, Traverso CE, Vagge A. Bilateral morphometric analysis of corneal sub-basal nerve plexus in patients undergoing unilateral cataract surgery: a preliminary in vivo confocal microscopy study. Br J Ophthalmol. 2021 Feb;105(2):174-179. doi: 10.1136/bjophthalmol-2019-315449. Epub 2020 Apr 3. PMID 32245849
- [Background] Guerrier, G., Abdoul, H., Jilet, L., Rothschild, P. R., Levy, J., Rondet, S., & Baillard, C. (2020). Musical intervention reduces anxiety-related hypertensive events during cataract surgery: A randomized controlled trial. Perioperative Care and Operating Room Management, 20, 100126. https://doi.org/10.1016/J.PCORM.2020.100126
- [Background] Guerrier G, Bernabei F, Lehmann M, Pellegrini M, Giannaccare G, Rothschild PR. Efficacy of Preoperative Music Intervention on Pain and Anxiety in Patients Undergoing Cataract Surgery. Front Pharmacol. 2021 Sep 30;12:748296. doi: 10.3389/fphar.2021.748296. eCollection 2021. PMID 34658886
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Harorani M, Davodabady F, Masmouei B, Barati N. The effect of progressive muscle relaxation on anxiety and sleep quality in burn patients: A randomized clinical trial. Burns. 2020 Aug;46(5):1107-1113. doi: 10.1016/j.burns.2019.11.021. Epub 2019 Dec 18. PMID 31862277
- [Background] Hashemi H, Pakzad R, Yekta A, Aghamirsalim M, Pakbin M, Ramin S, Khabazkhoob M. Global and regional prevalence of age-related cataract: a comprehensive systematic review and meta-analysis. Eye (Lond). 2020 Aug;34(8):1357-1370. doi: 10.1038/s41433-020-0806-3. Epub 2020 Feb 13. PMID 32055021
- [Background] Karwoski, B. A., Kazam, T. M. & Solomon, J. M. (2010). Music in the Operating Room and Patient Anxiety During Cataract Surgery. Invest. Ophthalmol. Vis. Sci, 51(13).
- [Background] Konopinska J, Lugowska D, Mariak Z, Obuchowska I. Comparison of auditory sensations in patients who underwent cataract phacoemulsification surgery in the first and second eye. Sci Rep. 2021 May 11;11(1):10026. doi: 10.1038/s41598-021-89594-6. PMID 33976341
- [Background] Lundstrom M, Dickman M, Henry Y, Manning S, Rosen P, Tassignon MJ, Young D, Behndig A, Stenevi U. Changing practice patterns in European cataract surgery as reflected in the European Registry of Quality Outcomes for Cataract and Refractive Surgery 2008 to 2017. J Cataract Refract Surg. 2021 Mar 1;47(3):373-378. doi: 10.1097/j.jcrs.0000000000000457. PMID 33086294
- [Background] Merakou K, Varouxi G, Barbouni A, Antoniadou E, Karageorgos G, Theodoridis D, Koutsouri A, Kourea-Kremastinou J. Blood Pressure and Heart Rate Alterations through Music in Patients Undergoing Cataract Surgery in Greece. Ophthalmol Eye Dis. 2015 Jun 11;7:7-12. doi: 10.4137/OED.S20960. eCollection 2015. PMID 26106264
- [Background] Mohammadpourhodki R, Sargolzaei MS, Basirinezhad MH. Evaluating the effect of massage based on slow stroke back massage on the anxiety of candidates for cataract surgery. Rom J Ophthalmol. 2019 Apr-Jun;63(2):146-152. PMID 31334393
- [Background] Mollaoğlu, M., Tuncay, F.Ö. ve Fertelli, T.K. (2011). İnmeli hasta bakım vericilerinde bakım yükü ve etkileyen faktörler. Dokuz Eylül Üniversitesi Hemşirelik Yüksekokulu Elektronik Dergisi, 3, 125-130.
- [Background] Molloy DW, Standish TI. A guide to the standardized Mini-Mental State Examination. Int Psychogeriatr. 1997;9 Suppl 1:87-94; discussion 143-50. doi: 10.1017/s1041610297004754. PMID 9447431
- [Background] Muddana SK, Hess OM, Sundar S, Venkatesh R. Preoperative and perioperative music to reduce anxiety during first-time phacoemulsification cataract surgery in the high-volume setting: randomized controlled trial. J Cataract Refract Surg. 2021 Apr 1;47(4):471-475. doi: 10.1097/j.jcrs.0000000000000485. PMID 33196574
- [Background] Musa A, Ng QX, Wai YZ, Iqbal T. Effect of slow tempo music on markers of anxiety during cataract surgery: Randomized control trial. Taiwan J Ophthalmol. 2021 Apr 30;12(1):74-81. doi: 10.4103/tjo.tjo_10_21. eCollection 2022 Jan-Mar. PMID 35399979
- [Background] Obuchowska I, Konopinska J. Fear and Anxiety Associated with Cataract Surgery Under Local Anesthesia in Adults: A Systematic Review. Psychol Res Behav Manag. 2021 Jun 18;14:781-793. doi: 10.2147/PRBM.S314214. eCollection 2021. PMID 34177276
- [Background] Öner, N. (2006). Türkiye'de Kullanılan Psikolojik Testlerden Örnekler. (2.Baskı). İstanbul: Boğaziçi Üniversitesi Yayınevi.
- [Background] Pager CK. Randomised controlled trial of preoperative information to improve satisfaction with cataract surgery. Br J Ophthalmol. 2005 Jan;89(1):10-3. doi: 10.1136/bjo.2004.048637. PMID 15615737
- [Background] Pellegrini M, Bernabei F, Schiavi C, Giannaccare G. Impact of cataract surgery on depression and cognitive function: Systematic review and meta-analysis. Clin Exp Ophthalmol. 2020 Jul;48(5):593-601. doi: 10.1111/ceo.13754. Epub 2020 Apr 20. PMID 32220125
- [Background] Socea SD, Abualhasan H, Magen O, Zayit-Soudry S, Blumenthal EZ, Duvdevan N, Mimouni M. Preoperative Anxiety Levels and Pain during Cataract Surgery. Curr Eye Res. 2020 Apr;45(4):471-476. doi: 10.1080/02713683.2019.1666996. Epub 2019 Sep 18. PMID 31509020
- [Background] Spielberger, C. D., Gonzalez-Reigosa, F., Martinez-Urrutia, A., Natalicio, L. F., & Natalicio, D. S. (2017). The State-Trait Anxiety Inventory. Revista Interamericana De Psicología/Interamerican Journal of Psychology, 5(3 & 4). https://doi.org/10.30849/rip/ijp.v5i3 & 4.620
- [Background] Wiwatwongwana D, Vichitvejpaisal P, Thaikruea L, Klaphajone J, Tantong A, Wiwatwongwana A; Medscape. The effect of music with and without binaural beat audio on operative anxiety in patients undergoing cataract surgery: a randomized controlled trial. Eye (Lond). 2016 Nov;30(11):1407-1414. doi: 10.1038/eye.2016.160. Epub 2016 Oct 14. PMID 27740618
- [Background] World Health Organization. (2021). Blindness and vision impairment. Https://Www.Who.Int/En/News-Room/Fact-Sheets/Detail/Blindness-and-Visual-Impairment Erişim tarihi 07.06.2022
- [Background] Yaman A, Buyukyilmaz F. The effect of relaxation exercises on burden, burnout, and anxiety levels in palliative caregivers. Perspect Psychiatr Care. 2022 Jul;58(3):1089-1095. doi: 10.1111/ppc.12906. Epub 2021 Jul 5. PMID 34227690
- [Background] Zemla AJ, Nowicka-Sauer K, Jarmoszewicz K, Wera K, Batkiewicz S, Pietrzykowska M. Measures of preoperative anxiety. Anaesthesiol Intensive Ther. 2019;51(1):64-69. doi: 10.5603/AIT.2019.0013. PMID 31280554